CLINICAL TRIAL: NCT07060391
Title: A Prospective Multicenter RCT Study of Deep Jugular Lymphovenous Anastomosis in the Treatment of Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yijun Cheng, Principal investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCLVA
Record Dates: First submitted 2025-06-22; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Experimental): Deep cervical lymphatic-venous anastomosis
  Interventions: Procedure: Deep cervical lymphatic-venous anastomosis
- Internal medicine conservative treatment (Placebo Comparator): Donepezil drug ,5-10mg,qd,po. All patients stopped taking cognitive-enhancing drugs and marketed therapeutic drugs such as ginkgo, high-dose vitamin E, lecithin, estrogen, non-steroidal anti-inflammatory drugs, Memegan, etc. after enrollment.
  Interventions: Drug: Donepezil drug treatment

INTERVENTIONS:
Procedure: Deep cervical lymphatic-venous anastomosis — Lymph node reconstruction was carried out using microsurgical techniques,improve cerebral lymphatic circulation and return, accelerate the excretion of pathological proteins, the metabolic products of the brain, from the brain. This is to delay the degenerative changes of the brain and the progression of Alzheimer's disease.
  Arms: Surgical treatment
Drug: Donepezil drug treatment — All patients stopped taking cognitive-enhancing drugs after enrollment, and marketed therapeutic drugs include ginkgo biloba, high-dose vitamin E, lecithin, estrogen, non-steroidal anti-inflammatory drugs, memegan, etc.
  Arms: Internal medicine conservative treatment

SUMMARY:
This research aims to observe the efficacy and safety of surgery compared with traditional medical treatment for moderate to severe dementia in Alzheimer's disease. This is a prospective multicenter RCT clinical research, involving a total of 3 research centers.Patients diagnosed with Alzheimer's disease accompanied by moderate to severe cognitive dysfunction in these three hospitals from January 2025 to January 2027 were included. This research is expected to recruit a total of 186 patients with moderate to severe Alzheimer's disease.93patients received conventional medical treatment, Deep cervical lymphatic-venous anastomosis was performed in 93 patients.Comprehensively evaluate the efficacy and safety of the patients within 48 weeks after treatment.

DETAILED DESCRIPTION:
Alzheimer's disease is a degenerative disorder of the central nervous system characterized by progressive cognitive dysfunction and behavioral impairment. At present, the treatment strategies for Alzheimer's disease include drug therapy, non-drug therapy and some emerging treatment methods. However, clinical evidence has confirmed that the effects of these treatment measures are limited. In recent years, Some neurosurgeons in China have begun to attempt to improve the disease progression of severe Alzheimer's disease through the innovative microscopic surgical method of deep jugular lymphovenous anastomosis. The therapeutic principle is Lymph node reconstruction is carried out using microsurgical techniques to improve the lymphatic circulation and return of the brain, accelerate the excretion of pathological proteins, the metabolic products of the brain, thereby delaying the degenerative changes of the brain and the progression of Alzheimer's disease. To verify the above assumption, this study will collaborate with a total of three institutions, namely Ruijin Hospital, Luwan Branch and Wuxi Branch. It is estimated that 186 patients with moderate to severe dementia of Alzheimer's disease will be included. They were randomly divided into the surgical treatment group (93 cases) and the traditional medical treatment group (93 cases). Cognitive function assessment, PETMR imaging examination, cerebrospinal fluid/blood testing and quality-adjusted life years were analyzed respectively at the 1st week, 4th week, 12th week, 24th week and 48th week after conservative treatment or surgery. To observe the efficacy and safety of surgery compared with traditional medical treatment for moderate to severe dementia in Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was clinically diagnosed with Alzheimer's disease and had a moderate to severe cognitive function score.
2. Age: 30-80 years old.
3. Gender is not limited.
4. The patient or their family members authorize their willingness to participate in this clinical trial and sign the informed consent form.
5. no contraindications for surgery.

Exclusion Criteria:

1. A history of radiotherapy or surgery for the head and neck.
2. Patients or their families with poor compliance who cannot strictly follow the rules.
3. Patients who cannot tolerate surgery.
4. Patients with other diseases that affect cognitive function.
5. Patients who cannot tolerate donepezil drug treatment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog score | baseline,48 weeks
  The improvement of 4 points by ADAS-cog is used as the judgment criterion for the clinical therapeutic effect, Compare the remission rates between the experimental group (surgery) and the control group (medication).

SECONDARY OUTCOMES:
Imaging data | From the first week to the 48th week
  PET-MRI labeled with specific tracers shows the changes in amyloid protein or tau deposition, Quantify and statistically analyze the changes between the two groups.
Cerebrospinal fluid examination | From the first week to the 48th week
  Test the Alzheimer's disease markers such as amyloid protein or tau deposition in the cerebrospinal fluid between the two groups, count the changes between the two groups.
Markers of Alzheimer's disease in the blood | From the first week to the 48th week
  Test the changes of Alzheimer's disease markers such as amyloid protein in the blood between the two groups,count the changes between the two groups.
Surgery-related adverse reactions | From the first week to the 48th week
  The occurrence of complications:such as postoperative bleeding,Peripheral nerve injury,Lymphatic vessel leakage,Cardiovascular and cerebrovascular events, etc.
Quality-Adjusted Life Year | From the first week to the 48th week
  It is a health outcome evaluation index that comprehensively considers survival time and quality of life. The survival time and quality of life of the intervention group and the medication group were compared. The calculation method is Survival Time (years) × Health Utility Value, The health utility value is a quality weight reflecting a specific health status(1 indicates complete health, 0 indicates death, and a negative value indicates a state worse than death). The utility values of patients under different health conditions were evaluated through the Quality of life assessment scale, an assessment should be conducted every six months after treatment. Multiply the duration of each health state by the corresponding utility value. Then accumulate to obtain the Quality-Adjusted Life Year score.

CONTACTS AND LOCATIONS:
Overall Officials: Yijun Cheng, Doc, Principal Investigator — Ruijin Hospital; Hanbing Shang, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No